CLINICAL TRIAL: NCT00985855
Title: Feasibility of Cetuximab (ERBITUX®) Associated With Concomitant Radio-chemotherapy in Patients With Locally Advanced Non Small Cell Lung Cancer: a Phase II, Randomised Study
Brief Title: Feasibility of Cetuximab Associated With Concomitant Radio-Chemotherapy in Patients With Locally Advanced Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-03; 2008-005013-21 (EudraCT Number)
Record Dates: First submitted 2009-09-22; First posted 2009-09-29 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2011-01

CONDITIONS: Non-Small-Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Cetuximab; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cisplatin, vinorelbine (Experimental): patients will receive induction chemotherapy (cisplatin, docetaxel) followed by a concomitant radio-chemothérapy including 2 cycles of cisplatin and vinorelbine associated with a weekly cetuximab infusion during the radiotherapy.
  Interventions: Drug: cisplatin, vinorlebine, cetuximab
- Cisplatin, etoposide (Experimental): patients will receive induction chemotherapy (cisplatin, docetaxel) followed by a concomitant radio-chemothérapy including 2 cycles of cisplatin and etoposide associated with a weekly cetuximab infusion during the radiotherapy.
  Interventions: Drug: cisplatine, etoposide, cetuximab

INTERVENTIONS:
Drug: cisplatin, vinorlebine, cetuximab — patient will receive 2 cycles of cisplatine 80 mg/m² at day 29 and day 50 more vinorelbine 15 mg/m² at day 29, day 36 and day 50 and 57 associated to cetuximab 400 mg/m² at day: 22,29, 36, 43, 50, 57, 64 and 71
  Arms: Cisplatin, vinorelbine
Drug: cisplatine, etoposide, cetuximab — patient will receive 2 cycles of cisplatine 50 mg/m² at day 29, 36, 57, and 64 + étoposide 50mg/m² during day 29-33, day 57-61associated to cetuximab 400 mg/m² at day: 22,29, 36, 43, 50, 57, 64 and 71
  Arms: Cisplatin, etoposide

SUMMARY:
Phase II, randomised, controlled, non comparative study with 2 parallel groups:

* Arm A: patients will receive induction chemotherapy (cisplatin and docetaxel) followed by a concomitant radio-chemotherapy including 2 cycles of cisplatin and vinorelbine associated with a weekly cetuximab infusion during the radiotherapy.
* Arm B: patients will receive induction chemotherapy (cisplatin and docetaxel) followed by a concomitant radio-chemothérapy including 2 cycles of cisplatin and etoposide associated with a weekly cetuximab infusion during the radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Non-Small-Cell Lung cancer cytologically or histologically proved
* Stage III AN2 inoperable or non resectable
* presence of at least one one dimension measurable target (at least 10 mm with spiral tomodensitometry)
* Possibility to include all targets in one irradiation field
* Age of 18 to 70
* Patients non previously treated
* Performance Status 0 or 1
* Loss of weight ≤10% in the 3 last months
* Neutrophil ≥ 1500/mm3 and platelets ≥ 100000/mm3
* Creatinine clearance ≥ 60 ml/min
* total bilirubin ≤ 1,5N and ASAT ALAT ≤ 2,5N
* Respiratory function normal: VEMS ≥ 40% theorical, DLCO/VA ≥ 50% theorical and PaO2 ≥ 60 mmHg
* Signed inform consent form
* Compliance to radiotherapy 66 Gy with dosimetry V20 ≤ 35% and pulmonary mean dose≤20 Gy

Exclusion Criteria:

* Pretreated bronchial carcinoma, excepted endoscopic deobstruction
* operable bronchial carcinoma
* small cell lung cancer, composite cancer, neuroendocrine cancer, broncho alveolar cancer
* superior vena cava syndroms
* puncturable pleural effusion
* metastatic lung cancer
* Stage IIIb cancer with neoplastic pericarditis
* Previous thoracic irradiation
* severe cardiac disease in the 12 months before inclusion
* interstitial lung disease
* anti-EGFR and anti-VEGF treatments
* hypersensitivity to murine proteins and allergies to protocol drugs
* uncontrolled infectious state
* HIV patient
* corticoid definitive contraindication
* péripheric neuropathy grade≥2
* neurologic, psychiatric and organic disorder
* past or concomitant cancer excepted treated skin baso-cellular cancer or in situ cervical cancer, or any cancer only surgically treated for 5 years
* breastfeeding woman

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
rate of patients presenting at least one toxicity grade≥3 (excepted hematological toxicity and nausea-vomiting) | End of concomitant treatment (Day 71)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre FOURNEL, Dr, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez, France